CLINICAL TRIAL: NCT01311778
Title: Cannabidiol as Treatment Intervention for Opioid Relapse
Brief Title: Study to Test the Safety and Efficacy of Cannabidiol as a Treatment Intervention for Opioid Relapse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hurd,Yasmin, Ph.D. (Individual)
Responsible Party: Principal Investigator, Yasmin Hurd, Principal Investigator, Hurd,Yasmin, Ph.D.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21DA027781 (NIH)
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Opiate Addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Cannabidiol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Subjects will receive placebo
  Interventions: Drug: Fentanyl
- CBD 400 mg (Experimental): Subjects will receive 400 mg CBD
  Interventions: Drug: Cannabidiol; Drug: Fentanyl
- CBD 800mg (Experimental): Subjects will receive 800 mg CBD
  Interventions: Drug: Cannabidiol; Drug: Fentanyl

INTERVENTIONS:
Drug: Cannabidiol — Subjects in Arm CBD 400 mg will receive 400 mg of Cannabidiol in two test sessions along with 0.5 mcg/kg and 1mcg/kg of fentanyl.
  Subjects in Arm CBD 800 mg will receive 800 mg of Cannabidiol in two test sessions along with 0.5 mcg/kg and 1mcg/kg of fentanyl.
  Arms: CBD 400 mg; CBD 800mg
Drug: Fentanyl — All subjects will receive 0.5 mcg/kg and 1mcg/kg of Fentanyl (test session 1 and test session 2)
  Other Names: Fentanyl Citrate

SUMMARY:
Despite the current available therapies for opioid-dependent patients, most patients relapse. This research project focuses on the development of a novel compound, cannabidiol, to modulate opioid craving in humans based on animal models showing its selective effectiveness to inhibit drug-seeking behavior. The development of a targeted treatment for opioid relapse would be of tremendous medical and public health value.

DETAILED DESCRIPTION:
Opioid abuse is a significant global public health problem. Of the over million opiate-dependent subjects today, only less than a quarter of such individuals receive treatment. Pharmacotherapeutic approaches traditionally have targeted 5 opioid receptors since heroin and its metabolites bind with highest affinity to this receptor subtype. Although such treatment strategies have improved substance abuse outcomes, they do not effectively block opiate craving and thus are still associated with high rates of relapse. Using a strategy of indirectly regulating neural systems to modulate opioid-related behavior, our preclinical rodent studies consistently demonstrated that cannabidiol (CBD), a nonpsychoactive component of cannabis, specifically inhibited cue- induced heroin-seeking behavior. CBD's selective effect on drug-seeking behavior was pronounced after 24 hrs and endured even two weeks after the last drug administration following short-term CBD exposure. The fact that drug craving is generally triggered by exposure to conditioned cues suggests that CBD might be an effective treatment for heroin craving, specially given its protracted impact on behavior. CBD has already been shown in various clinical studies to be well tolerated with a wide safety margin in human subjects. CBD thus represents a strong candidate for the development as a potential therapeutic agent in humans for opioid craving and relapse prevention. It is the goal of this exploratory phase of the project to (1) determine the safety and basic pharmacokinetic characteristics of CBD when administered concomitantly with opiate in humans and (2) characterize the acute (24 hr) and short-term (3 days) effects of CBD administration on cue-induced craving in drug-abstinent heroin-dependent subjects using a random double blind design. This exploratory investigation together with ongoing complementary preclinical rodent studies has the potential to significantly impact the development of a novel agent for drug relapse prevention that is critical for ending the continued cycle of substance abuse. PUBLIC HEALTH RELEVANCE: Despite the current available therapies for opioid-dependent patients, most patients relapse. This research project focuses on the development of a novel compound, cannabidiol, to modulate opioid craving in humans based on animal models showing its selective effectiveness to inhibit drug-seeking behavior. The development of a targeted treatment for opioid relapse would be of tremendous medical and public health value.

ELIGIBILITY:
Inclusion Criteria:

* being aged between 21 and 65 years old.
* having exposure at least once to an opioid (i.e. codeine, morphine, Fentanyl) in the past

Exclusion Criteria:

* using any psychoactive drug or medication at any time during the study, or 24 hours before the test session
* having a past or current diagnosis of drug abuse or dependence (except for nicotine), based on the SCID-IV interview (Structured Clinical Interview for DSM-IV)
* being maintained on methadone or buprenorphine, or taking opioid antagonist such as naltrexone
* having taken any opioid in the last 14 days
* having medical conditions, including Axis I psychiatric conditions under DSM-IV (examined with the MINI International Neuropsychiatric Interview-MINI), history of cardiac disease, arrhythmias, head trauma, and seizures
* having a history of hypersensitivity to any opioid or cannabinoid
* being pregnant or breastfeeding
* not using an appropriate method of contraception such as hormonal contraception (oral hormonal contraceptives, Depo-Provera, Nuva-Ring), intrauterine device (IUD), sterilization, or double barrier method (combination of any two barrier methods used simultaneously, i.e. spermicide, diaphragm)
* arriving to the study site visibly intoxicated as determined by a clinical evaluation for signs and symptoms of intoxication and as verified by a drug screen for cocaine, cannabis, opiates, benzodiazepines, barbiturates, phencyclidine and amphetamines
* being actively treated and currently involved in an addiction treatment program
* being an anesthesiologist or a pharmacist

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety of cannabidiol oral administration prior to fentanyl IV administration. | 9 timepoints: -10 min, 30, 60, 90, 120, 180, 240, 360, 480
  We will assess safety and adverse effects with the Systematic Assessment for Treatment Emergent Events (SAFTEE). Excessive sedation (GCS<10), cardiac dysrhythmia (on telematry monitor), hypotension (blood pressure < 90/60 mmHg), bradycardia (heart rate 50/minute),severe anxiety, or seizures (partial or generalized tonic-clonic) after the administration of either Fentanyl or Cannabidiol would result in discontinuation of the study for the subject and immediate medical attention.

SECONDARY OUTCOMES:
General cannabidiol pharmacokinetics | 9 timepoints: -10 min, 30, 60, 90, 120, 180, 240, 360, 480
  Blood will be taken at specified times to determine cannabidiol peak plasma concentration (Cmax), time to reach peak serum concentration (tmax) and serum elimination half-life (t1/2).
Cortisol levels | -10 min, 30, 60, 90, 120, 180, 240, 360, 480
  Variation in plasma levels of cortisol will be measured at various time points.
Cannabidiol clearance | 5 timepoints: -60 min, 45, 120, 240, 480
  Urine will be taken at specified times to estimate cannabidiol concentration in order to assess clearance and excretion functions.
Vital signs-BP | -10, 30, 60, 75, 90, 120, 180, 240, 360, 480 min
  Blood pressure (mmHg) will be monitored and change from baseline will be studied across the multiple time points.
Vital signs-HR | -10, 30, 60, 75, 90, 120, 180, 240, 360, 480 min
  Heart rate (beats/minute) will be monitored and change from baseline will be studied across the multiple time points.
Vital signs - RR | -10, 30, 60, 75, 90, 120, 180, 240, 360, 480 min
  respiratory rate (respirations/minute) will be monitored and change from baseline will be studied across the multiple time points.
Vital signs - O2 | -10, 30, 60, 75, 90, 120, 180, 240, 360, 480 min
  % oxygen saturation will be monitored and change from baseline will be studied across the multiple time points.
Vital signs - temp | -10, 30, 60, 75, 90, 120, 180, 240, 360, 480 min
  body temperature (degrees Fahrenheit) will be monitored and change from baseline will be studied across the multiple time points.
Vital signs - EKG | -10, 30, 60, 75, 90, 120, 180, 240, 360, 480 min
  EKG will be monitored and change from baseline will be studied across the multiple time points.
Subjective measures-VAS | -1, 30, 65, 90, 120, 240, 360, 480 min.
  Questionnaires will be used to measure subjective responses. Anxiety will be assessed using a visual analog scale (VAS).
Subjective measures-PANAS | -1, 30, 65, 90, 120, 240, 360, 480 min.
  Questionnaires will be used to measure subjective responses. The PANAS (Positive and Negative Affect Schedule) will allow obtaining positive and negative affect measures.
Subjective measures-Opiate effect | -1, 30, 65, 90, 120, 240, 360, 480 min.
  Questionnaires will be used to measure subjective responses. Global Intoxication and Withdrawal Rating will be administered to assess potential variations in the subjective effects associated to fentanyl.
Subjective measures- OVAS | -1, 30, 65, 90, 120, 240, 360, 480 min.
  Questionnaires will be used to measure subjective responses. Opiate Visual Analog Scales (OVAS) will be administered to assess potential variations in the subjective effects associated to fentanyl.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hurd, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States